CLINICAL TRIAL: NCT03863860
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Multicenter Trial of Maintenance Treatment With Fluzoparib Capsules Versus Placebo in Patients With Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: A Trial of Maintenance Treatment With Fluzoparib Versus Placebo in Relapsed Ovarian Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FZPL-Ⅲ-301-OC
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluzoparib capsules, 50mg per capsule (Experimental): Fluzoparib capsules, PO
  Interventions: Drug: Fluzoparib capsules
- Placebo capsules, 50mg per capsule (Placebo Comparator): Placebo capsules, PO
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Fluzoparib capsules — Fluzoparib capsules
  Other Names: SHR-3162
  Arms: Fluzoparib capsules, 50mg per capsule
Drug: Placebo capsules — Placebo capsule
  Other Names: Placebo
  Arms: Placebo capsules, 50mg per capsule

SUMMARY:
To evaluate the efficacy, safety tolerability of maintenance therapy with Fluzoparib(A PARP inhibitor) versus placebo in Chinese patients with recurrent ovarian cancer who achieved a complete response (CR) or partial response (PR) after platinum-based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed high-grade serous or endometrioid ovarian cancer (including primary peritoneal and fallopian tube cancer)
2. Completion of ≥2 previous platinum-containing regimens
3. Complete response (CR) or partial response (PR) achieved with last platinum-based chemotherapy regimen as determined by investigator
4. Ability to be randomized ≤8 weeks after last dose of platinum

Exclusion Criteria:

1. Prior treatment with a poly (ADP-ribose) polymerase (PARP) inhibitor
2. Patients who have received other study drug treatment within 4 weeks prior to the first administration(< 5 elimination half-lives of the study drug molecular targeted anti-cancer drugs).
3. Patients with clinical symptoms of cancer ascites, pleural effusion, who need to drainage, or who have undergone ascites drainage within 2 months prior to the first administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Progression free survival(PFS) by Blinded Independent Review Committee (BIRC) in relapsed ovarian cancer patients | up to 2 years
  Defined as progression free survival per RECIST 1.1 criteria
Progression free survival(PFS) by BIRC in relapsed ovarian cancer patients with Breast cancer susceptibility gene(BRCA) mutant | up to 2 years
  Defined as progression free survival per RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression free survival(PFS) in relapsed ovarian cancer patients | up to 2 years
  PFS is Progression-Free-Survival per RECIST 1.1 criteria
Time to progression(TTP) by Gynecological Cancer Intergroup(GCIG) CA 125 criteria | up to 2 years
  TTP is Time to Progression
Chemotherapy free interval (CFI) CFI | up to 2 years
  CFI is the time from last platinum dose until initiation of next anticancer therapy (excluding maintenance therapy if used following the penultimate regimen)
overall survival(OS) | up to 3 years
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up
Objective Response Rate | At baseline,at the time point of every 12 weeks, up to 2 years
  Objective Response Rate complete or partial response per RECIST 1.1 criteria
Adverse Events(AEs) and Serious Adverse Events (SAEs) | from the first drug administration to within 30 days for the last treatment dose
  assess the safety and tolerability of Fluzoparib maintenance monotherapy in platinum sensitive relapsed ovarian cancer patients by record the number of Participants with of AEs and SAEs, and the proportion of patients with AEs and SAEs, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li N, Zhang Y, Wang J, Zhu J, Wang L, Wu X, Yao D, Wu Q, Liu J, Tang J, Yin R, Lou G, An R, Zhang G, Xia X, Li Q, Zhu Y, Zheng H, Yang X, Hu Y, Zhang X, Hao M, Huang Y, Lin Z, Wang D, Guo X, Yao S, Wan X, Zhou H, Yao L, Yang X, Cui H, Meng Y, Zhang S, Qu J, Zhang B, Zou J, Wu L. Fuzuloparib Maintenance Therapy in Patients With Platinum-Sensitive, Recurrent Ovarian Carcinoma (FZOCUS-2): A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Trial. J Clin Oncol. 2022 Aug 1;40(22):2436-2446. doi: 10.1200/JCO.21.01511. Epub 2022 Apr 11. PMID 35404684